CLINICAL TRIAL: NCT05196698
Title: Home High Flow Oxygen to Reduce Acute Exacerbation of COPD
Acronym: HIFAE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019/0412/HP
Record Dates: First submitted 2021-11-30; First posted 2022-01-19 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Flow Oxygen Therapy (Experimental)
  Interventions: Other: High Flow Oxygen Therapy
- Long-Term Oxygen Therapy (Other): Control arm
  Interventions: Other: Long-term oxygen therapy

INTERVENTIONS:
Other: High Flow Oxygen Therapy — HFOT will be delivered validated medical devices and established as follow:
  * Patient will be acclimatized to HFOT which will aim to achieve a flow of air of 30L/min at a temperature of 34°C using dedicated nasal canula.
  * Once patient acclimatized, oxygen will be entrained in the HFOT device at a flow that will aim to achieve a saturation > 90%. An arterial blood gas will be performed with such oxygen delivery, flowrate and temperature to ensure a PaO2 ≥ 8kPa
  Arms: High Flow Oxygen Therapy
Other: Long-term oxygen therapy — LTOT delivery will be performed according to French guidelines
  Arms: Long-Term Oxygen Therapy

SUMMARY:
The objective of the study is to evaluate the efficacy of home High Flow Oxygen for the reduction of severe exacerbation following admission for a severe exacerbation of COPD or death against standard oxygen therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with a diagnosis of COPD defined by GOLD guidelines
2. Admitted in hospital for AECOPD
3. With severe respiratory impairment defined by one of the following criteria (long-term oxygen therapy (LTOT) criteria):

   * Previously established on long-term oxygen therapy according to the following criteria: PaO2 < 7.3kPa or <8kPa with polycythemia, pulmonary hypertension or right heart failure on room air in stable condition Or
   * PaO2 < 7.3kPa or <8kPa with polycythemia, pulmonary hypertension or right heart failure on room air after clinical stabilization during the index admission
4. Patients affiliated or, beneficiary of a social security cover
5. Patient who has read and understood the information letter and signed the consent form
6. For woman of childbearing potential, use of an effective contraception (oestro-progestatives or intra-uterine device or tubal ligation) since at least 1 month and an blood pregnancy test by β-HCG negative at the screening visit, during the duration of the study
7. For menopausal woman: confirmatory diagnosis (amenorrhea not medically induced for at least 12 months before the inclusion visit)

Exclusion Criteria:

1. Age <18 or > 85 years
2. Patient treated with chronic NIV with ongoing treatment
3. Patients diagnosed with obstructive sleep apnea (OSA) treated with CPAP. Diagnosis of OSA will be over-ruled in patient that had a previous overnight polygraphy. For patients who never had an overnight polygraphy, screening for OSA will be made using the STOP-BANG questionnaire. If the results of the STOP-BANG questionnaire (Appendix 1) is >3, an Apnea-link recording will be performed. If AHI>30/h, patient will be excluded.
4. BMI > 35 kg/m2
5. Patient admitted for an acute COVID-19 infection
6. Hypercapnic respiratory failure justifying NIV defined as

   1. An Arterial Blood Gas (ABG) PaCO2 > 7 kPa in stable condition within 6 months
   2. Patients with ABG PaCO2 > 7 kPa at hospital discharge and that remained hypercapnic between 2- and 4-weeks following discharge
7. Pregnancy (blood pregnancy test positive) or lactation ongoing
8. Significant psychiatric disorder or dementia that would prevent adherence to study protocol
9. Tobacco use < 10 pack-year
10. Expected survival < 12 months due to any situation other than COPD disease
11. Refusal of high-flow oxygen therapy
12. Person deprived of liberty by administrative or judicial decision or placed under judicial protection (guardianship or supervision)
13. Patients already involved in a research protocol that would impact with the outcome measured in the current protocol

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Estimated)
Dates: Start 2022-08-26 (Actual); Primary Completion 2026-08-26 (Estimated); Study Completion 2026-08-26 (Estimated)

PRIMARY OUTCOMES:
time to first hospital admission for Acute Exacerbation of Chronic Obstructive Pulmonary Disease | 12 months
time to death | 12 months

SECONDARY OUTCOMES:
Change from Baseline in Health-related Quality of Life | 3 months
  Health-related quality of life is evaluated using Saint-Georges Respiratory score
Change from Baseline in Health-related Quality of Life | 6 months
  Health-related quality of life is evaluated using Saint-Georges Respiratory score
Change from Baseline in Health-related Quality of Life | 12 months
  Health-related quality of life is evaluated using Saint-Georges Respiratory score
Change from Baseline in Health-related Quality of Life | 3 months
  Health-related quality of life is evaluated using EuroQol-5D-5L score
Change from Baseline in Health-related Quality of Life | 6 months
  Health-related quality of life is evaluated using EuroQol-5D-5L score
Change from Baseline in Health-related Quality of Life | 12 months
  Health-related quality of life is evaluated using EuroQol-5D-5L score
Change from Baseline in Health-related Quality of Life | 3 months
  Health-related quality of life is evaluated using Hospital anxiety and depression scale
Change from Baseline in Health-related Quality of Life | 6 months
  Health-related quality of life is evaluated using Hospital anxiety and depression scale
Change from Baseline in Health-related Quality of Life | 12 months
  Health-related quality of life is evaluated using Hospital anxiety and depression scale
Change from Baseline in Health-related Quality of Life | 3 months
  Health-related quality of life is evaluated using Leicester Cough Questionnaire score
Change from Baseline in Health-related Quality of Life | 6 months
  Health-related quality of life is evaluated using Leicester Cough Questionnaire score
Change from Baseline in Health-related Quality of Life | 12 months
  Health-related quality of life is evaluated using Leicester Cough Questionnaire score
Change from Baseline in Health-related Quality of Life | 3 months
  Health-related quality of life is evaluated using Chronic Obstructive Pulmonary Disease Assessments Test score
Change from Baseline in Health-related Quality of Life | 6 months
  Health-related quality of life is evaluated using Chronic Obstructive Pulmonary Disease Assessments Test score
Change from Baseline in Health-related Quality of Life | 12 months
  Health-related quality of life is evaluated using Chronic Obstructive Pulmonary Disease Assessments Test score
Change from Baseline in Health-related Quality of Life | 3 months
  Health-related quality of life is evaluated using Pittsburgh sleep quality index score
Change from Baseline in Health-related Quality of Life | 6 months
  Health-related quality of life is evaluated using Pittsburgh sleep quality index score
Change from Baseline in Health-related Quality of Life | 12 months
  Health-related quality of life is evaluated using Pittsburgh sleep quality index score
Number of Adverse events | 3 months
  Imputability of Adverse events is evaluated by investigator
Number of Adverse events | 6 months
  Imputability of Adverse events is evaluated by investigator
Number of Adverse events | 12 months
  Imputability of Adverse events is evaluated by investigator

CONTACTS AND LOCATIONS:
Overall Officials: Antoine CUVELIER, Pr, Principal Investigator — University Hospital, Rouen; Maxime PATOUT, Dr, Principal Investigator — AP-HP La Pitié Salpétrière
Locations (1):
- UHRouen, Rouen, France

IPD SHARING:
Plan to Share IPD: No